CLINICAL TRIAL: NCT02453061
Title: A Comparative Phase 2 Study Assessing the Efficacy of Triheptanoin, an Anaplerotic Therapy in Huntington's Disease
Acronym: TRIHEP3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C14-62
Record Dates: First submitted 2015-05-12; First posted 2015-05-25 (Estimated); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — triheptanoin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo group (Placebo Comparator): Subjects will receive safflower oil at 1g/kg/day for 6 months (months 0 - 6) and triheptanoin oil at 1g/kg/day for 6 months (months 7 - 12)
  Interventions: Drug: Placebo
- Triheptanoin group (Active Comparator): Subjects will receive triheptanoin oil at 1g/kg/day for 6 months (months 0 - 6) and triheptanoin oil at 1g/kg/day for 6 months (months 7 - 12)
  Interventions: Drug: Triheptanoin oil

INTERVENTIONS:
Drug: Triheptanoin oil — Triheptanoin oil orally administered at 1g/kg/day
  Arms: Triheptanoin group
Drug: Placebo — Safflower oil orally administered at 1g/kg/day
  Arms: Placebo group

SUMMARY:
In the study the investigators plan to include 100 early affected HD patients (5 ≤ UHDRS ≤ 40) in a randomized, double-blind, controlled study in 2 centers (France and the Netherlands). Patients will receive either triheptanoin at 1g/kg of body weight per day (n = 50), or a control oil (n = 50) at 1g/kg of body weight per day for 6 months followed by an open label phase using triheptanoin for another 6 months. Efficacy of triheptanoin will be evaluated by measurements of caudate volume using volumetric magnetic resonance imaging. Clinical improvement will be evaluated by brain energy metabolism quantification as evaluated by the ratio of inorganic phosphate/phosphocreatine, during visual stimulation, using 31P-MRS, UHDRS, TFC, and PBA-S scores as well as performance on the neuropsychological battery. Patient quality of life will be evaluated with the SF-36 questionnaire before and after treatment; biological tolerance and compliance will be evaluated by routine biochemical blood tests, plasma and urine measurements of triheptanoin oil derivatives and patient report.

ELIGIBILITY:
Inclusion Criteria:

* Positive genetic test with CAG repeat length ≥39 in HTT gene
* At least 18 years of age
* Signature of informed consent
* Covered by social security
* UHDRS score between 5 and 40
* Ability to undergo MRI scanning
* BMI between 18 and 30

Exclusion Criteria:

* Hypersensitivity to triheptanoin or to one of its excipients
* Additional major comorbidities
* History of severe head injury
* Participation in another therapeutic trial (3 month exclusion period)
* For women of childbearing age, the absence of two forms of effective contraception (with the exception of those who are abstinent)
* Pregnancy or breastfeeding
* Inability to understand information about the protocol
* Persons deprived of their liberty by judicial or administrative decision
* Adult subject under legal protection or unable to consent
* Treatment with tetrabenazine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
volumetric magnetic resonance imaging | 6 months
  A decrease in the rate of caudate atrophy, using volumetric MRI

SECONDARY OUTCOMES:
motor function after 6 months | 6 months
  Decrease in the progression of the UHDRS United Huntington's Disease Rating Scale after 6 months of treatment
31- Phosphorus Magnetic Resonance Spectroscopy | 3 months
  An increase in the index of brain energy restoration - as defined by the difference between Pi/PCr ration during visual stimulation and the mean of the Pi/PCr ratio during rest and recovery - using 31P-MRS
Caudal Atrophy | 12 months
  Rate of caudate atrophy, using volumetric MRI
motor function after 12 months | 12 months
  Decrease in the progression of the UHDRS United Huntington's Disease Rating Scale after 12 months of treatment
Patient autonomy after 6 months | 6 months
  Stability of the Total Functional Capacity (TFC) after 6 months of treatment
Patient autonomy after 12 months | 12 months
  Stability of the Total Functional Capacity (TFC) after 12 months of treatment
Sustained restoration of brain energy metabolism after 6 months | 6 months
  Sustained restoration of brain energy metabolism using 31P-MRS after 6 months of treatment
Sustained restoration of brain energy metabolism after 12 months | 12 months
  Sustained restoration of brain energy metabolism using 31P-MRS after 12 months of treatment
Symbol Digit Modalities Test after 6 months | 6 months
  The benefit of triheptanoin on cognitive function will be evaluated after 6 months using a neuropsychological battery including the SDMT (Symbol Digit Modalities Test), a test of visuomotor coordination
Symbol Digit Modalities Test after 12 months | 12 months
  The benefit of triheptanoin on cognitive function will be evaluated after 12 months using a neuropsychological battery including the SDMT (Symbol Digit Modalities Test), a test of visuomotor coordination
Stroop test after 6 months | 6 months
  The benefit of triheptanoin on cognitive function will be evaluated after 6 months using a neuropsychological battery including the Stroop test, a test evaluating concentration and capacity for inhibition
Stroop test after 12 months | 12 months
  The benefit of triheptanoin on cognitive function will be evaluated after 12 months using a neuropsychological battery including the Stroop test, a test evaluating concentration and capacity for inhibition
Trail making test after 6 months | 6 months
  The benefit of triheptanoin on cognitive function will be evaluated after 6 months using a neuropsychological battery including the Trail making test, a test to evaluate mental flexibility
Trail making test after 12 months | 12 months
  The benefit of triheptanoin on cognitive function will be evaluated after 12 months using a neuropsychological battery including the Trail making test, a test to evaluate mental flexibility
Digit span test after 6 months | 6 months
  The benefit of triheptanoin on cognitive function will be evaluated after 6 months using a neuropsychological battery including the Digit span test, a test evaluating attention and working memory
Digit span test after 12 months | 12 months
  The benefit of triheptanoin on cognitive function will be evaluated after 12 months using a neuropsychological battery including the Digit span test, a test evaluating attention and working memory
psychiatric symptoms after 3 months | 3 months
  The effect of triheptanoin on psychiatric symptoms will be evaluated after 3 months with the PBA-S, an evaluation of problem behaviors associated with HD
psychiatric symptoms after 6 months | 6 months
  The effect of triheptanoin on psychiatric symptoms will be evaluated after 6 months with the PBA-S, an evaluation of problem behaviors associated with HD
psychiatric symptoms after 9 months | 9 months
  The effect of triheptanoin on psychiatric symptoms will be evaluated after 9 months with the PBA-S, an evaluation of problem behaviors associated with HD
psychiatric symptoms after 12 months | 12 months
  The effect of triheptanoin on psychiatric symptoms will be evaluated after 12 months with the PBA-S, an evaluation of problem behaviors associated with HD
patients' daily life | 6 months
  The global impact of triheptanoin on patients' daily life will be evaluated at the end of the blinded treatment period using qualitative research methods. To statistically test whether experts classify treated and not treated patients better than could be expected by chance, a permutation test based on a modified version of Fisher's Lady tasting tea procedure will be used (Fischer 1935).
quality of life questionnaire after 6 months | 6 months
  A standardized quality of life questionnaire, the Short Form-36 Health Survey, will be used after 6 months
quality of life questionnaire after 12 months | 12 months
  A standardized quality of life questionnaire, the Short Form-36 Health Survey, will be used after 12 months
Number of adverse events | 12 months
  Safety of triheptanoin will be evaluated based on review of adverse events
clinical exam for Long term tolerance | 12 months
  Long-term tolerance will be confirmed by clinical exam at study visits
home nurse visits for Long term tolerance | 12 months
  Long-term tolerance will be confirmed by patient report during home nurse visits

CONTACTS AND LOCATIONS:
Locations (2):
- Département de Génétique, Paris, France
- Department of Neurology, Leiden, Netherlands

REFERENCES:
- [Derived] Mochel F, Meneret A, Adanyeguh IM, Giron C, Hainque E, Luton MP, Atencio M, Debs R, Jacobs M, Veldkamp FCM, Barbier M, Coppen EM, van der Zwaan KF, Diallo A, Ottolenghi C, Vicaut E, Roos RA, Durr A. Effect of Triheptanoin on Caudate Atrophy and Motor Scores in Patients With Early-Stage Huntington Disease: A Phase II Study. Neurology. 2025 Jan 28;104(2):e210194. doi: 10.1212/WNL.0000000000210194. Epub 2024 Dec 30. PMID 39804569
- [Derived] Rodrigues FB, Ferreira JJ, Wild EJ. Huntington's Disease Clinical Trials Corner: June 2019. J Huntingtons Dis. 2019;8(3):363-371. doi: 10.3233/JHD-199003. PMID 31381524

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT02453061/SAP_001.pdf